CLINICAL TRIAL: NCT02874625
Title: Randomized Clinical Trial in Children to Evaluate the Biocompatibility of Resin-based Dental Materials
Brief Title: RCT to Evaluate Biocompatibility of Resin-based Dental Materials
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: S57169
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Materials Testing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment 1 (Active Comparator): Dental restoration performed with glass-ionomer materials.
  Interventions: Procedure: Dental restoration
- Treatment 2 (Experimental): Dental restoration performed with resin-based composites.
  Interventions: Procedure: Dental restoration

INTERVENTIONS:
Procedure: Dental restoration — Teeth with caries will be restored

SUMMARY:
In this randomized clinical trial, the bio-compatibility of 2 materials used for dental restorations will be compared: glass-ionomer vs resin-based composites.

Urine and saliva samples will be taken for determination of bisphenol A levels at several time points, and for analysis of the estrogenic activity using ERE-CALUX.

Also buccal cells will be taken. Next, DNA extraction will be done with a commercial kit. Global alterations in DNA methylation and DNA hydroxymethylation levels will be determined using UPLC-MS/MS.

ELIGIBILITY:
Inclusion Criteria:

* one or more carious lesions in primary molars that require treatment

Exclusion Criteria:

* carious lesions that already affected the dental pulp, large lesions requiring cusp replacement, presence of oral inflammatory conditions during the previous 2 weeks, carriage of a fixed or removable prosthesis/orthodontic appliance, chronic disease requiring intake of drugs, exposure to diagnostic X-rays in previous 2 months, previous dental restorations

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2017-08-30 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Urinary bisphenol A levels | 1 year
Salivary bisphenol A levels | 1 year
%DNA methylation | 6 months
%DNA hydroxymethylation | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- BIOMAT, Department of Oral Health Sciences, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No